CLINICAL TRIAL: NCT02694835
Title: Initial Performance of a Modified Daily Disposable Silicone Hydrogel Contact Lens
Brief Title: Initial Performance of a Modified Daily Disposable Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CLP691-C001
Record Dates: First submitted 2016-02-12; First posted 2016-03-01 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-02

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- DT1 UV (Experimental): Delefilcon A contact lenses with Ultraviolet (UV) Absorber worn bilaterally (in both eyes) for 9 hours
  Interventions: Device: Delefilcon A contact lenses with UV Absorber
- DT1 (Active Comparator): Delefilcon A contact lenses worn bilaterally for 9 hours
  Interventions: Device: Delefilcon A contact lenses

INTERVENTIONS:
Device: Delefilcon A contact lenses with UV Absorber
  Other Names: DAILIES TOTAL1® UV (DT1 UV)
  Arms: DT1 UV
Device: Delefilcon A contact lenses
  Other Names: DAILIES TOTAL1® (DT1)
  Arms: DT1

SUMMARY:
The purpose of this study is to evaluate the incidence of ocular discomfort device-related adverse events with DAILIES TOTAL1® with UV Absorber (DT1 UV) contact lenses compared with current DAILIES TOTAL1® (DT1) contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an Informed Consent document;
* Current wearers of commercial DT1 lenses (for at least 3 months), with a minimum wearing time of 5 days per week and 8 hours per day;
* Spherical contact lens correction within the range of -2.00 to -4.00 Diopter (D) in both eyes;
* Manifest astigmatism less than or equal to 0.75 D (at screening);
* Best-corrected visual acuity (BCVA) greater than or equal to 20/25 in each eye (as determined by manifest refraction at screening);
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Eye injury in either eye within 12 weeks prior to study enrollment;
* Any anterior segment infection, inflammation, disease, or abnormality that contraindicates contact lens wear as determined by the Investigator;
* Use of systemic or ocular medications for which contact lens wear could be contraindicated, including topical ocular medications and lubrication drops that would require instillation during contact lens wear;
* History of herpetic keratitis;
* History of refractive surgery or irregular cornea;
* Pathologically dry eye that precludes contact lens wear;
* Concurrent participation (or within the previous 30 days) in a contact lens or lens care product clinical trial;
* Monocular (only 1 eye with functional vision);
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2016-04-11 (Actual); Study Completion 2016-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, GCRA, Study Director — Alcon Research

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 5 investigational sites located in the United States.
Pre-assignment Details: Of the 81 enrolled, 1 subject exited as a screen failure prior to randomization. This reporting group includes all randomized subjects (80).
Groups:
- Dailies Total1 (DT1): Delefilcon A contact lenses worn bilaterally for 9 hours
Period: Overall Study
Arm/Group | DT1 UV | Dailies Total1 (DT1)
Started (Randomized and Treated) | 41 | 39
Completed | 41 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects who were exposed to the investigational product and satisfied specific evaluability criteria (Full Analysis Set).
Groups:
- Total: Total of all reporting groups
Arm/Group | DT1 UV | Dailies Total1 (DT1) | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (8.5) | 35.3 (9.9) | 35.8 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 23 | 57
  Male | 7 | 16 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 36 | 35 | 71
  Black or African American | 2 | 0 | 2
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Island | 0 | 0 | 0
  Multi-Racial | 0 | 0 | 0
  Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidence (Number) of Ocular Discomfort Device-related Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a subject who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. Reported in units of eyes.
Time Frame: Day 1 at Hour 9 ± 3 hours
Population: Full Analysis Set
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | DT1 UV | Dailies Total1 (DT1)
Number analyzed (Participants) | 41 | 39
Number analyzed (Eyes) | 82 | 78
Eyes | 0 | 0

ADVERSE EVENTS:
Time Frame: Duration of enrollment = 1 Day
Description: AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol. This analysis population includes all subjects/eyes exposed to any investigational product evaluated in the study.
Arm/Group | DT1 UV | Dailies Total1 (DT1)
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/39
Other Adverse Events (participants affected / at risk) | 0/41 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.